CLINICAL TRIAL: NCT05821062
Title: Effect of Antiplatelet Therapies in Patients With Depression and Coronary Disease
Brief Title: Antiplatelet Therapies in Patients With Depression and Coronary Disease
Acronym: ENHANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1422
Record Dates: First submitted 2023-03-08; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Depression
Keywords: Coronary Artery Disease; Depression; Acetylsalicylic acid; Prasugrel; Ticagrelor; Dual antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease; Depression | interventions — Clopidogrel; cysteine and glycine-rich protein 3; Therapeutics; Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — platelet activation, coagulation, lipid peroxidation, CLP active metabolite and epigenetic modifications influencing the response to CLP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Group 1a: CAD patients with depression on standard ASA+CLP therapy.
  Interventions: Other: standard Aspirin (ASA) + clopidogrel (CLP) therapy
- Group 1b: CAD Patients without depression on standard ASA+CLP therapy.
  Interventions: Other: standard Aspirin (ASA) + clopidogrel (CLP) therapy
- Group 2a: CAD patients with depression on standard ASA+TCG/PSG therapy.
  Interventions: Other: standard Aspirin (ASA) + Ticagrelor (TCG) or Prasugrel (PSG) therapy
- Group 2b: CAD patients without depression on standard ASA+TCG/PSG therapy.
  Interventions: Other: standard Aspirin (ASA) + Ticagrelor (TCG) or Prasugrel (PSG) therapy
- Group 3a: CAD patients with depression on standard ASA treatment alone at least 1 month after TCG/PSG cessation.
  Interventions: Other: standard ASA therapy
- Group 3b: CAD patients without depression on standard ASA treatment alone at least 1 month after TCG/PSG cessation.
  Interventions: Other: standard ASA therapy
- Group 1c: Subjects with depression without CAD (DS) are enrolled are enrolled as a comparison group.
- Group 1d: Healthy control subjects (HC), subjects without depression and without CAD are enrolled as a comparison group.

INTERVENTIONS:
Other: standard Aspirin (ASA) + clopidogrel (CLP) therapy — ASA100mg + CLP 75mg daily
  Groups: Group 1a; Group 1b
Other: standard Aspirin (ASA) + Ticagrelor (TCG) or Prasugrel (PSG) therapy — ASA 100 mg + TCG 90mg/b.i.d or PSG10mg daily
  Groups: Group 2a; Group 2b
Other: standard ASA therapy — ASA 100 mg daily
  Groups: Group 3a; Group 3b

SUMMARY:
Depression after an acute coronary syndrome (ACS) but also at any time after CAD diagnosis, is highly associated with death, and it predicts mortality more than any other risk factor, comorbidity or follow-up events, suggesting that the standard medical therapy may not be sufficient to prevent the poor prognosis in these patients.

This study aims to assess whether depression might affect the response to dual antiplatelet therapy (DAPT) as recommended in coronary artery disease (CAD) patients.

Specific aims:

* to evaluate whether depression affects the antithrombotic response during Aspirin (ASA) plus clopidogrel (CLP) therapy in CAD patients.
* to assess the antithrombotic effects of ASA plus ticagrelor or prasugrel (TCG/PSG) therapy in CAD patients with depression by evaluating pro-thrombotic phenotype in CAD patients with and without depression during ASA+TCG/PSG.
* to assess whether there is or not the reactivation of pro-thrombotic profile after cessation of dual antiplatelet therapy in CAD patients with or without depression in single antiplatelet therapy after TCG/PSG cessation.

DETAILED DESCRIPTION:
This study is a multicentre, prospective, observational, case-control, and cross-sectional study. It is planned to enrol 400 patients/subjects (300 patients at Centro Cardiologico Monzino and 100 subjects at IRCCS National Neurological Institute "C. Mondino" Foundation).

Pharmacological treatments in progress will be recorded, administration of Beck Depression Inventory-II (BDI-II), and a fasting blood venous sample (from ante-cubital vein) will be carried out for the haematochemical analyses and for research samples. First morning-urine will be collected for oxidative stress evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Centro Cardiologico Monzino: Patients/subjects of both sexes, aged between 18 and 85 years with or without depression, with CAD:

   * Group 1: CAD patients in ASA+CLP (100mg+75mg/daily) therapy with the absence of acute coronary symptoms for at least 5 months.
   * Group 2: CAD patients in ASA+TCG/PSG (TCG:90mg/b.i.d or PSG:10mg/daily) therapy, at least 6 months after ACS.
   * Group 3: CAD patients during ASA treatment alone at least 1 month after TCG/PSG cessation.
2. IRCCS National Neurological Institute "C. Mondino" Foundation:

   * Group 1: Patients/subjects of both sexes, aged between 18 and 85 years with or without depression, without CAD.

Exclusion Criteria:

* severe chronic heart failure (NYHA class III/IV)
* severe concomitant valvular disease
* infectious pathologies
* autoimmune diseases
* haematological diseases
* serious kidney or liver failure
* positive anamnesis for current or previous neoplasia in the 5 years prior to enrolment
* positive anamnesis for major traumas and/or surgery in the 6 months prior to enrolment
* taking immunosuppressive drugs
* taking of anti-inflammatory drugs
* taking of antidepressant drugs
* presence of dementia and psychiatric disorders other than depression
* Coronavirus disease-19 (COVID-19) swab positive

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study includes patients/subjects with or without depression, with CAD (to be enrolled at Centro Cardiologico Monzino) and without CAD (to be enrolled at IRCCS National Neurological Institute "C. Mondino" Foundation)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Verify whether depression affects the platelet response during ASA plus CLP therapy in CAD patients | 3 years
  Measuring platelet activity markers
Verify whether depression affects the coagulation during ASA plus CLP therapy in CAD patients | 3 years
  Measuring all the parameters of clot formation and lysis collected by thromboelastography analyses
Verify whether depression affects oxidative stress during ASA plus CLP therapy in CAD patients | 3 years
  Measuring lipid peroxidation
Assess the effects of ASA plus TCG/PSG therapy on platelet response in CAD patients with depression | 3 years
  Measuring platelet activity markers
Assess the effects of ASA plus TCG/PSG therapy on coagulation in CAD patients with depression | 3 years
  Measuring all the parameters of clot formation and lysis collected by thromboelastography analyses
Assess the effects of ASA plus TCG/PSG therapy on oxidative stress in CAD patients with depression | 3 years
  Measuring lipid peroxidation
Assess whether there is or not the activation of platelet response after cessation of dual antiplatelet therapy in CAD patients with depression | 3 years
  Measuring platelet activity markers
Assess whether there is or not the activation of coagulation after cessation of dual antiplatelet therapy in CAD patients with depression | 3 years
  Measuring all the parameters of clot formation and lysis collected by thromboelastography analyses
Assess whether there is or not the activation of oxidative stress after cessation of dual antiplatelet therapy in CAD patients with depression | 3 years
  Measuring lipid peroxidation

SECONDARY OUTCOMES:
CLP metabolism in patients with depression and CAD | 3 years
  Measuring the CLP active metabolite
Epigenetic modification in patients with depression and CAD | 3 years
  Through miRNAs analysis
DNA methylation in patients with depression and CAD | 3 years
  Measuring DNA methylation levels of two 5'-C-phosphate-G-3' (CpG) dinucleotides on P2Y12
Impact of depression on oxidative stress in patients without CAD | 3 years
  Measuring platelet activity markers
Effect of depression on oxidative stress in patients without CAD | 3 years
  Measuring lipid peroxidation

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Marenzi, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (2):
- Italy (2):
  - IRCCS Centro Cardiologico Monzino, Milan
  - IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia